CLINICAL TRIAL: NCT02017080
Title: Efficacy Of Non Invasive Diagnostic Procedures In Evaluating The Influence Of Maternal Autoimmune Thyroid Gland Disease On Fetus
Brief Title: Fetal Thyroid Ultrasound And Fetal Thyroid Hormones
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Svetlana Spremovic Radjenovic, Assistant professor, Gynecologyst and Obstetrician, sibspecialist in endocrinology, University of Belgrade
Other Study IDs: 440/VI-3
Record Dates: First submitted 2013-12-15; First posted 2013-12-20 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Pregnancy Complicated by Hyperthyroidism; Hypothyroidism in Pregnancy
Keywords: fetal thyroid ultrasound; fetal fT4; antithyroid antibodies; pregnancy; autoimmune thyroid disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hyperthyroid pregnant women: Autoimmune hyperthyroidism diagnosed and treated by an endocrinologist, based on clinical and laboratory tests and ultrasound clinical examination
- Hypothyroid pregnant women: Autoimmune hypothyroidism diagnosed and treated by an endocrinologist, based on clinical and laboratory tests and ultrasound thyroid examination
- Healthy pregnant women: Euthyroid women with uncomplicated pregnancies, with antithyroid antibodies within reference ranges

SUMMARY:
Non invasive methods: maternal antithyroid antibodies and ultrasound measurement of the fetal thyroid gland could be an important tool for detecting fetal thyroid dysfunction in mothers with autoimmune thyroid disease.

DETAILED DESCRIPTION:
Autoimmune thyroid disease complicates 5-20% unselected pregnancies. The crucial impacting factor on the pregnancy outcomes in mothers with autoimmune thyroid disease is the thyroxine level changes.

But, fetal hypo or hyperthyroidism can be found in treated pregnant women with autoimmune thyroid disease, even when their thyroid hormones are in normal range, because thyroid antibodies, antithyroid drugs and iodine pass the placenta.

Our previous results show that high fetal free thyroxine (fT4) levels measured by cordocentesis are unexpectedly frequent in women with autoimmune thyroid disease, including maternal autoimmune hypo- and hyperthyroidism. Increasing awareness that even some mild fetal disorder can have an impact on later neurophysiologic development and the health of an individual makes the recognition and therapy of fetal hypo- or hyperthyroidism an increasingly significant domain of interest. According to our results, fetal fT4 concentrations did not correlate neither with dose of medication nor with ultrasound biometric parameters; the range for maternal thyroid-stimulating hormone (TSH) correlated predominantly with normal fT4 can not be marked off. The type and concentration of antithyroid antibodies might have some prognostic value.

There is a growing list of publications referring to the ultrasound measurement of the fetal thyroid as an important tool for detecting fetal thyroid dysfunction. Fetal thyroid measurement became a part of the clinical guidelines for pregnancies complicated with maternal thyroid disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed and treated for autoimmune hyper or hypothyroidism: - Disease diagnosed by an endocrinologist, based on clinical and laboratory tests and ultrasound thyroid examination.
* All of the hyper or hypothyroid women have to be positive for one or both thyroid antibodies when entering the study.
* Patients with autoimmune thyroid disease will be included into the study in the first half of pregnancy, but not later than 20th weeks of gestation
* For the pregnant women in control group:
* if they are euthyroid, with antithyroid antibodies within reference range, healthy and have uncomplicated pregnancy

Exclusion Criteria:

* Patients with chronic diseases (except for thyroid disease) in their past medical history record. Pregnancy induced diseases are not a part of the exclusion criteria (gestational diabetes and pregnancy induced hypertension)
* all the patients whose pregnancies resulted from assisted reproductive technologies will be excluded from the study.
* mothers from the control group will be excluded, if the neonate have abnormal thyroid function

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Groups are selected from State tertiary referral centre for Gynecology and Obstetrics
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Fetal thyroid size measured by ultrasonography | 28th week of gestation

SECONDARY OUTCOMES:
Fetal fT4 | 28th week of gestation
  Sampled at the same time when fetal thyroid measurement is done
Fetal antithyroid antibodies | 28th week of gestation
  Fetal antithyroid antibodies: thyroid peroxidase (TPO), TSH receptor (TRAK), thyroglobuline (Tg) antibodies, will be measure in the same sample as fetal fT4
Maternal fT4 | 28th week of gestation
  Sampled at the same time as the fetal free thyroxin and fetal antithyroid antibodies
Maternal TSH | 28th week of gestation
  Measured in the same sample as maternal fT4
Maternal antithyroid antibodies | 28th week of gestation
  Measured in the same sample as maternal fT4 Maternal antithyroid antibodies: thyroid peroxidase (TPO), TSH receptor (TRAK), thyroglobuline (Tg) antibodies, will be measured in the same sample as fetal fT4

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana S Spremovic- Radjenovic, MD PhD, Principal Investigator — Medical School of the University of Belgrade
Locations (1):
- Clinic for Gynecology and Obstetrics , Clinical Center of Serbia, Belgrade, Serbia

REFERENCES:
- [Background] Achiron R, Rotstein Z, Lipitz S, Karasik A, Seidman DS. The development of the foetal thyroid: in utero ultrasonographic measurements. Clin Endocrinol (Oxf). 1998 Mar;48(3):259-64. doi: 10.1046/j.1365-2265.1998.00388.x. PMID 9578813
- [Background] Ranzini AC, Ananth CV, Smulian JC, Kung M, Limbachia A, Vintzileos AM. Ultrasonography of the fetal thyroid: nomograms based on biparietal diameter and gestational age. J Ultrasound Med. 2001 Jun;20(6):613-7. doi: 10.7863/jum.2001.20.6.613. PMID 11400935
- [Result] Luton D, Le Gac I, Vuillard E, Castanet M, Guibourdenche J, Noel M, Toubert ME, Leger J, Boissinot C, Schlageter MH, Garel C, Tebeka B, Oury JF, Czernichow P, Polak M. Management of Graves' disease during pregnancy: the key role of fetal thyroid gland monitoring. J Clin Endocrinol Metab. 2005 Nov;90(11):6093-8. doi: 10.1210/jc.2004-2555. Epub 2005 Aug 23. PMID 16118343